CLINICAL TRIAL: NCT02955888
Title: A Phase 2, Double-Blind, Placebo Controlled Study to Evaluate the Safety & Tolerability of PBI-4050 and Its Effects on Pancreatic and Pulmonary Function in Cystic Fibrosis Patients With Abnormal Glucose Tolerance
Brief Title: Study of Safety, Tolerability & Efficacy in Cystic Fibrosis Patients With Abnormal Glucose Tolerance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unsatisfactory rate of recruitment
Sponsor: Liminal BioSciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBI-4050-CT-9-07
Record Dates: First submitted 2016-10-21; First posted 2016-11-04 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — setogepram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBI4050 (Experimental): Four 200 mg capsules (total 800 mg) administered orally, once daily.
  Interventions: Drug: PBI4050
- Placebo (Placebo Comparator): Four 200 mg capsules (total 800 mg) administered orally, once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBI4050 — Investigational Medicinal Product
  Arms: PBI4050
Drug: Placebo — Comparator
  Arms: Placebo

SUMMARY:
This is a Phase 2, multi-center, double blind, placebo controlled study to evaluate the safety and tolerability of PBI-4050, and its effects on the pancreatic, pulmonary functions and on various biomarkers in Cystic Fibrosis patients with abnormal glucose tolerance. Patients with abnormal glucose tolerance have elevated glucose level either at 1 hour or 2 hour during an Oral Glucose Tolerance Test (OGTT). The Main study will include 24 weeks of treatment with PBI-4050 or matching placebo. At the end of the treatment period, patients will have the option of participating in a 24-week Extension study.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, double blind, placebo controlled study to evaluate the safety and tolerability of PBI-4050, and its effects on the pancreatic, pulmonary functions and on various biomarkers in Cystic Fibrosis patients with abnormal glucose tolerance. Patients with abnormal glucose tolerance have elevated glucose level either at 1 hour or 2 hour during an Oral Glucose Tolerance Test (OGTT).

A total of 90 patients will be enrolled for study participation. A Data Safety Monitoring Board (DSMB) will continually review individual patients safety data obtained from the 90 patients. When the first 15 patients have completed at least 1 month of study treatment, the DSMB will meet formally to determine whether additional patients may be enrolled, the study should continue with changes or if the study should be stopped. In addition, the DSMB will review the PK data and may recommend dose adjustment based on the PK results.

The total duration of study participation for each patient is at least 32 weeks, including up to 4 weeks of a screening period, 24 weeks of study treatment and 4 weeks of safety follow-up.

Patients who choose to participate in the open label extension will be in the study for an additional 24 weeks of study treatment and 4 weeks of safety follow-up (for a total of 56 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older at screening.
2. Patient has a documented and confirmed CF diagnosis.
3. Patient has performed an OGTT for diagnosis of INDENT, IGT and de novo CFRD within 12 months prior to screening visit.
4. Patient has a Body Mass Index (BMI) of at least 17 kg/m2.
5. Patient has signed written informed consent.
6. Patient is able and willing to self-monitor blood glucose level at home.
7. Female patients of childbearing potential must have a negative pregnancy test (serum or urine) and agree to use adequate birth control from screening throughout the study and for the 30 days after the last study drug administration.
8. If a male patient has not been vasectomized at least 6 months before screening and partners with a woman of childbearing potential, he must be willing to use an acceptable contraceptive method throughout the study and for the 30 days after the last study drug administration.

Exclusion Criteria:

1. Patient has recent or ongoing infection requiring intravenous treatment with an anti-infective agent within 30 days before screening.
2. Patient is concurrently taking high dose of ibuprofen (>30 mg/kg) or is using corticosteroids (except inhaled and topical corticosteroids).
3. Patient is currently using weight-loss medications.
4. 4. Patient has used any moderate/potent inhibitor of cytochrome P450 (CYP) 2C9 isozyme or strong inhibitor of CYP3A isozyme within 30 days prior to the first study drug administration.
5. Patient has significantly elevated liver enzyme levels, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 Upper Limit of Normal (ULN) or total bilirubin above ULN at screening.
6. Patient has a history of chronic alcohol or other substance abuse as determined at screening that may prevent study compliance based on Investigator judgment.
7. History of malignancy of any organ system, treated or untreated, within the past 5 years other than basal or squamous cell skin cancer.
8. Patient has unstable chronic heart failure that has required change in therapy within 2 months prior to screening.
9. Patient with known non-controlled history of infection with Human Immunodeficiency Virus (HIV) and/or active Hepatitis.
10. Woman who is pregnant, breast-feeding or planning a pregnancy during the course of the study.
11. Woman of childbearing potential who is unwilling to use adequate birth control throughout the duration of the study.
12. Patient has any condition that, in the Investigator's opinion, is likely to interfere with study conduct and compliance.
13. Patient has participated in an investigational clinical trial within 30 days (or 5 half-lives, whichever is longer) prior to screening visit.
14. Patient is under insulin and/or repaglinide treatment at screening/baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events (Combined Main Study and Extension Study Participation) | Baseline to 1 Year
  Adverse Event data (including abnormal laboratory values) collected up to final follow-up (30 days after last dose of study drug). Serious Adverse Events that were ongoing at the follow-up visit will be followed until the event resolved, returned to baseline, or was determined to be a stable or chronic condition.

SECONDARY OUTCOMES:
Change from Baseline in glucose level following Oral Glucose Tolerance Test (OGTT) (Combined Main Study and Extension Study Participation) | Up to 1 Year
Change from Baseline of insulin-secretion following Oral Glucose Tolerance Test (OGTT) (Combined Main Study and Extension Study Participation) | Up 1 Year
Change from Baseline of HbA1C following Oral Glucose Tolerance Test (OGTT) (Combined Main Study and Extension Study Participation) | Up to 1 Year
Change from Baseline in pulmonary function parameters (FEV1 ) (Combined Main Study and Extension Study Participation) | Up to 1 Year
Change from Baseline in pulmonary function parameters ( FVC) (Combined Main Study and Extension Study Participation) | Up to 1 Year
Change from Baseline in pulmonary function parameters (FEV1/FVC ratio) (Combined Main Study and Extension Study Participation) | Up to 1 Year
Change from Baseline in pulmonary function parameters (Forced Expiratory Flow (FEF25%-75%)) (Combined Main Study and Extension Study Participation) | Up to 1 Year
Change from baseline in weight (Combined Main Study and Extension Study Participation) | Up to1 Year

OTHER OUTCOMES:
Changes from baseline in fibrotic and inflammatory biomarkers in blood (Combined Main Study and Extension Study Participation) | Up to 1 Year
Changes from baseline in fibrotic and inflammatory biomarkers in urine (Combined Main Study and Extension Study Participation) | Up to1 Year

CONTACTS AND LOCATIONS:
Overall Officials: John Moran, MD, Study Chair — Liminal BioSciences Ltd.
Locations (7):
- Canada (7):
  - St. Paul's Hospital - Pacific Lung Health Centre (PLHC), Vancouver, British Columbia
  - Queen Elizabeth II Health Science Center, Halifax, Nova Scotia
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de Recherches Cliniques de Montréal (IRCM), Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de l'Université Laval (IUCPQ), Québec

IPD SHARING:
Plan to Share IPD: No